CLINICAL TRIAL: NCT02190396
Title: Vitamin D Deficiency and Placental Calcification in Low-risk Obstetric Population - Are They Related?
Status: Completed | Type: Observational
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Ali Ozgur Ersoy, Medical Doctor, Zekai Tahir Burak Women's Health Research and Education Hospital
Other Study IDs: VIT D PLACENTAL CALCIFICATION
Record Dates: First submitted 2014-06-21; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: Vitamin D Deficiency
Keywords: Calcium; Vitamin D; Placental calcification.
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Maternal venous and umbilical cordon blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Group 1: Placental calcification of Grade 3
- Group 2: No placental calcification noted, the control group.

SUMMARY:
Maternal vitamin D deficiency has been suggested to influence fetal and neonatal health. The role of placenta in vitamin D regulation is known but alteration of Vitamin D levels at placental pathologies is unknown. Placental calcification is usually thought to be a physiological aging process. Nevertheless, it can be a pathological change resulting from the effects of environmental factors on the placenta. The aim of the investigators study was to evaluate the relationship between placental calcification and maternal and cord blood 25-hydroxyvitamin-D3 [25(OH)D] and calcium concentrations in low-risk obstetric population at term and their consequences.

DETAILED DESCRIPTION:
Vitamin D deficiency is a public health problem prevalent throughout the World. Low blood 25-hydroxyvitamin D3 ( 25OHD ) level was found to be associated with preeclampsia, gestational diabetes, infectious diseases, decrease in fetal bone mineralization, and increase in fetal respiratory infections and infant wheezing [1].

Requirement of vitamin D is primarily met by the exposure of skin to sun and secondarily by intake of food. The provision of vitamin D from the skin depends upon melanin pigment, the use of sun screens, age, dressing style and seasonal changes [1]. Placenta plays an important role in Vitamin D metabolism during pregnancy and some independent risk factors increasing the risk of placental dysfunction at fetomaternal interface also influence vitamin D metabolism [2,3]. Nevertheless, there can be a pathological change resulting from the effects of environmental factors on the placenta .

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy

Exclusion Criteria:

* Foreknown systemic diseases, multiple pregnancy, smoking cigarettes, receiving vitamin D or calcium supplementation.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who admitted our clinic without foreknown systemic diseases or multiple pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with low birth weight. | Three months

SECONDARY OUTCOMES:
Percentage of delivery with cesarean section. | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Ali O Ersoy, Principal Investigator — Medical doctor
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Wuertz C, Gilbert P, Baier W, Kunz C. Cross-sectional study of factors that influence the 25-hydroxyvitamin D status in pregnant women and in cord blood in Germany. Br J Nutr. 2013 Nov;110(10):1895-902. doi: 10.1017/S0007114513001438. Epub 2013 May 23. PMID 23697742
- [Background] Cho GJ, Hong SC, Oh MJ, Kim HJ. Vitamin D deficiency in gestational diabetes mellitus and the role of the placenta. Am J Obstet Gynecol. 2013 Dec;209(6):560.e1-8. doi: 10.1016/j.ajog.2013.08.015. Epub 2013 Aug 14. PMID 23954530
- [Background] Saffery R, Ellis J, Morley R. A convergent model for placental dysfunction encompassing combined sub-optimal one-carbon donor and vitamin D bioavailability. Med Hypotheses. 2009 Dec;73(6):1023-8. doi: 10.1016/j.mehy.2009.03.057. Epub 2009 Oct 9. PMID 19819084